CLINICAL TRIAL: NCT00858559
Title: Follow-up of Patients With Implantable Cardioverter Defibrillators by Home Monitoring (ANVITE)
Acronym: ANVITE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped due to low enrollment. Patients will be followed up for 3 months.
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HS047
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2011-05

CONDITIONS: Cardiac Pacing; Electric Countershock; Ventricular Tachyarrhythmia
Keywords: Implantable cardioverter defibrillator; Remote monitoring; Follow-up
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Home Monitoring
  Interventions: Device: Implantable cardioverter defibrillator with Home Monitoring function
- 2 (Active Comparator): Home Monitoring not used
  Interventions: Device: Standard implantable cardioverter defibrillator

INTERVENTIONS:
Device: Implantable cardioverter defibrillator with Home Monitoring function — Implantable cardioverter defibrillators can send data from its diagnostic and therapy memory via wireless Home Monitoring on a daily basis to an internet based platform, securely accessed by the attending physician
  Other Names: Lumax 500/540 VR-T; CardioMessenger (for Home Monitoring data transmission)
  Arms: 1
Device: Standard implantable cardioverter defibrillator — Implantable cardioverter defibrillators used as standard devices without Home Monitoring
  Other Names: Lumax 500/540 VR-T
  Arms: 2

SUMMARY:
Patients with implantable cardioverter defibrillators (ICDs) should undergo regular device follow-ups every 3 months, to verify proper ICD function. However, many follow-ups are uneventful, revealing no relevant changes related to the implanted device and in the patient's diagnostic and therapeutic status. For time and economic reasons, longer follow-up intervals are frequently used although they are not according to recommendations. This may increase the delay in detection of relevant changes in the disease and in deviations from optimal ICD therapy in the individual patients. In the newest ICDs, the essential parameters reflecting safety and appropriateness of ICD therapy (threshold, impedance, intracardiac electrogram, etc.) are transmitted via Home Monitoring on a daily basis, to an internet platform accessible by the attending physician.

In the present study, the investigators evaluate safety and efficacy of 12-month follow-up intervals in ICDs with Home Monitoring capability, as compared with conventional 3-month follow-up scheme.

ELIGIBILITY:
Inclusion Criteria:

* Indication for a single-chamber implantable cardioverter-defibrillator (ICD)

Exclusion Criteria:

* Contraindication for ICD
* Indication for dual-chamber ICD or cardiac resynchronization therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-03; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Significant adverse events, especially death, hospitalization, inadequate device therapies | 27 months

SECONDARY OUTCOMES:
All-cause mortality | 27 months
Number of device follow-ups | 27 months
Quality of life | 27 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Perings, M.D., Principal Investigator — Cardiology in Tangram House, Düsseldorf, Germany
Locations (1):
- Cardiology in Tangram House, Düsseldorf, Germany